CLINICAL TRIAL: NCT02507830
Title: Mesh Fixation With a Synthetic Glue in Primary Inguinal Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Meshg2
Record Dates: First submitted 2015-07-20; First posted 2015-07-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glubran 2 fixation: Mesh fixation with Glubran 2 glue in primary inguinal hernia repair

SUMMARY:
Prospective observational study with mesh fixation using FDA approved synthetic glue,glubran 2 and standard mesh fixation with stiches in primary inguinal hernia repair surgery. The investigators aim is to recruit 150 patients for the study.

The outcomes The investigators would like to determine are : postoperative pain,recurrences and complication rates such as seromas.

DETAILED DESCRIPTION:
Prospective observational study with mesh fixation using FDA approved synthetic glue,glubran 2 and standard mesh fixation with stiches in primary inguinal hernia repair surgery. The investigators aim is to recruit 150 patients for the study.

The outcomes The investigators would like to determine are : postoperative pain,recurrences and complication rates such as seromas.

ELIGIBILITY:
Inclusion Criteria:

* Primary Inguinal hernia

Exclusion Criteria:

* Recurrent hernia
* Large inguinoscrotal hernias
* Bilateral inguinal hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults older than 18 undergoing a primary inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain (Evaluation will be conducted through scale and a questionnaire ) | 2 years

SECONDARY OUTCOMES:
Hernia recurrence (Evaluation will be conducted through a questionnaire and physical examination ) | 2 years
Postoperative complications (Evaluation will be conducted through a questionnaire and physical examination ) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Adel Abu_Salih, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel